CLINICAL TRIAL: NCT05720585
Title: Intervention of Mobile Health Application for Older Adults With Subjective Memory Complaints
Brief Title: Subjective Memory Complaints' Cognitive Intervention
Acronym: SMCCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hongli Chen (Other)
Responsible Party: Sponsor-Investigator, Hongli Chen, Research assistant, Nanjing Medical University
Organization: Nanjing Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NMU-IRB-(2019)437
Record Dates: First submitted 2022-12-11; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-01

CONDITIONS: Subjective Memory Complaint

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental)
  Interventions: Other: Intervention of mobile health application

INTERVENTIONS:
Other: Intervention of mobile health application — According to the contents of the Subjective Memory Complaint (SMC) application intervention program for the older adults previously formulated, the intervention time and the frequency (30min / time, once a week) of each training module and other contents were determined. The application will be implemented and lasted for a total of 1 month.

SUMMARY:
This study will be divided into two parts: development of the mobile medical application for older adults with subjective memory decline and the intervention application. Start by developing and optimizing the application based on the rapid prototyping model. Then, in accordance with the framework of designing and evaluating complex intervention measures proposed by the Medical Research Council of the United Kingdom, pre-experiments will be carried out to apply the developed application to the actual intervention process to test the intervention effect, feasibility, and other contents of the application.

ELIGIBILITY:
Inclusion Criteria:

* Patients with subjective memory complaints by SMCQ for 6 months and above.
* Individuals age over 60 years (depending on the characteristics of the disease, it can be relaxed to 55 years) are included.
* Older adults owning and being able to use smartphones to access the Internet, or whose caregivers can assist in the completion can also be included.
* Older adults who voluntary participate in the study and provide informed consent are also included.

Exclusion Criteria:

* Older adults diagnosed with cognitive or mild cognitive impairment.
* Older adults diagnosed with other neurological disorders ( cerebrovascular disease, encephalitis, brain tumor, brain trauma, epilepsy, Parkinson 's disease, depression, mania, etc. ), metabolic diseases ( anemia, thyroid dysfunction, folic acid and vitamin B12 deficiency, etc. ), carbon monoxide poisoning and cognitive decline caused by general anesthesia
* Older adults with serious medical and surgical diseases who cannot complete the experiment are also excluded.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-02-15 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Subjective Memory Complaint (SMC) | Change from Baseline Subjective Memory Complaint at 1 month
  Subjective Memory Complaint Questionnaire (SMCQ), a SMC self-assessment questionnaire designed for the elderly population, is adopted. There are 14 items in 2 dimensions. The first 4 items are used to evaluate the overall memory and the last 10 items are used to evaluate the daily memory.
Cognitive Function | Change from Baseline Cognitive function at 1 month
  Montreal Cognitive Assessment (MoCA) is adopted, which includes 8 aspects of cognitive domain assessment. The total score of this scale is 30 points, the higher the score is, the better the cognitive function will be. .
Memory | Change from Baseline Memory at 1 month
  The Auditory Verbal Learning Test (AVLT), developed by Kwak in 2001, is used to test the verbal memory function of the older adults.
The Quality of Life Rating Scale (SF-12) | Change from Baseline Quality of Life at 1 month
  The Quality of Life Rating Scale (SF-12) is used. There are 12 items in total, with 8 dimensions, which are general health, physiological function, physiological function, physical pain, mental health, vitality, social function and emotional function. The eight dimensions can be summarized into two comprehensive indicators of physical health and mental health.

SECONDARY OUTCOMES:
Demographic characteristics | Base line
  General demographic of the older adults with memory complaints are obtained by self-made questionnaires including age, gender, education, occupation, whether they live alone, and chronic diseases.

IPD SHARING:
Plan to Share IPD: No